CLINICAL TRIAL: NCT04334187
Title: Feasibility and Accessibility of a Mindfulness-based Smoking Cessation Intervention for NYCHA Residents
Brief Title: NYCHA Mindfulness-based Smoking Cessation Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the pandemic's impacts on being able to conduct the intervention for this study, unable to begin recruitment.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-01435
Record Dates: First submitted 2020-03-26; First posted 2020-04-06 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smoke Cessation Group (Experimental): Mindfulness-based smoking cessation sessions will follow the mindfulness based addiction treatment (MBAT) intervention for smoking cessation. Sessions are in group format for two hours, weekly. Two groups of sessions with about 10 participants per group will be organized.
  Interventions: Behavioral: Mindfulness Based addition treatment

INTERVENTIONS:
Behavioral: Mindfulness Based addition treatment — The intervention is comprised of 8 weekly group MBAT sessions. Two weekly groups of about 10 participants each will be conducted. All participants will also have the option to receive nicotine patches, gum, or lozenges for four weeks as part of their time in the study. Participants will complete surveys at enrollment (baseline), immediately after their last MBAT session (around 2 months after enrollment) and one month after completing treatment (3 months post-enrollment). Surveys will assess primary and secondary outcomes and satisfaction with the intervention.

SUMMARY:
The study will assess feasibility, accessibility and impact of a mindfulness-based smoking cessation group intervention for New York City Housing Authority (NYCHA) residents. Residents who smoke to receive an 8-week intervention. Participants will also be offered 4 weeks of nicotine replacement therapy (NRT).

DETAILED DESCRIPTION:
The primary objective of this research is to examine the feasibility, accessibility and impact of a mindfulness-based smoking cessation program for NYCHA residents.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Current smoker (>= 5 cigarettes per day). Dual tobacco users are eligible as long as their primary tobacco product is cigarettes.
* Ready to quit smoking cigarettes within 30 days
* Able to attend the 8 weekly MBAT sessions at the scheduled days/times
* NYCHA resident
* English language
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Patient Health Questionnaire-2 (PHQ-2) score indicating current risk for depression
* Self-reported diagnosis of schizophrenia, bipolar disorder, schizotypal disorder or other psychotic disorder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who perceive the Mindfulness based addiction treatment as useful at time of Enrollment | Baseline
  Participants will report their perceived usefulness and effectiveness of the intervention using self reported surveys at enrollment (baseline).
Number of participants who perceive the Mindfulness based addiction treatment as useful after last MBAT session. | 2 months
  Number of participants will report their perceived usefulness and effectiveness of the intervention using self reported surveys after their last MBAT session (2 months after enrollment).
Number of participants who perceive the Mindfulness based addiction treatment as useful post treatment | 3 months
  Participants will report their perceived usefulness and effectiveness of the intervention using self reported surveys one month after completing treatment (3 months post-enrollment).
Number of participants who perceive the Mindfulness based addiction treatment as effective | 3 months
  Participants who self-report 7-day abstinence in the final follow up survey (3 months) will provide a biochemically validated saliva sample

SECONDARY OUTCOMES:
Number of participants who adhered to the Mindfulness based addiction treatment | 3 months
  This will be reported in the number of sessions attended and completed mindfulness exercises in between the sessions.
Number of participants who self reported abstinence | 2 months
  This will be self reported at the end of the treatment (2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rogers, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Erin.rogers@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.